CLINICAL TRIAL: NCT01098357
Title: A Phase I/II, Multicentre, Randomised, Controlled, and Open-label Trial Comparing the Efficacy and Safety of Three Dose Regimens of BioChaperone PDGF-BB to Becaplermin Gel for the Treatment of Diabetic Foot Ulcer
Brief Title: Comparative Study of 3 Dose Regimens of BioChaperone to Becaplermin Gel for the Treatment of Diabetic Foot Ulcer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Virchow Group (Industry)
Collaborators: Adocia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC1-CT1
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2012-08

CONDITIONS: Diabetic Foot Ulcers
Keywords: rhPDGF, diabetic foot ulcer,
MeSH Terms: conditions — Diabetic Foot | interventions — Becaplermin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Biochaperone PDGF-BB low dose (Experimental): BioChaperone PDGF-BB is a new formulation of the B isoform dimer of recombinant human Platelet-Derived Growth Factor (rhPDGF-BB) containing the new excipient Biochaperone, a dextran modified polymer. The finished product is a sterile multi-dose spray vial.
  Interventions: Drug: Biochaperone PDGF-BB Low dose
- Biochaperone PDGF-BB High dose (Experimental): BioChaperone PDGF-BB is a new formulation of the B isoform dimer of recombinant human Platelet-Derived Growth Factor (rhPDGF-BB) containing the new excipient Biochaperone, a dextran modified polymer. The finished product is a sterile multi-dose spray vial.
  Interventions: Drug: Biochaperone PDGF-BB High dose
- Regranex (Active Comparator): Becaplermin gel (Regranex® Gel 0.01%, Systagenix, formerly and Johnson & Johnson) is a topical gel of rhPDGF-BB conditioned in a gel tube.
  Interventions: Drug: Regranex
- Very Low Dose BioChaperone PDGF-BB (Experimental): BioChaperone PDGF-BB Very Low Dose sprayed on the wound every two days (e.g., Mondays, Wednesdays and Fridays) for 20 weeks or until complete wound healing, at the dose of 4 µg/cm²/application
  Interventions: Drug: Biochaperone PDGF-BB Very Low Dose

INTERVENTIONS:
Drug: Biochaperone PDGF-BB Low dose — BioChaperone PDGF-BB low dose is applied as a spray every two days at the dose of 12.5 µg/cm2 for up to 20 weeks
  Other Names: BC low dose
  Arms: Biochaperone PDGF-BB low dose
Drug: Biochaperone PDGF-BB High dose — BioChaperone PDGF-BB high dose is applied as a spray every two days at the dose of 25 µg/cm2 for up to 20 weeks
  Other Names: BC high dose
  Arms: Biochaperone PDGF-BB High dose
Drug: Regranex — Regranex gel is applied once daily at the dose of 6.25 µg/cm2 for up to 20 weeks
  Other Names: Becaplermin
  Arms: Regranex
Drug: Biochaperone PDGF-BB Very Low Dose — BioChaperone PDGF-BB Very Low Dose sprayed on the wound every two days (e.g., Mondays, Wednesdays and Fridays) for 20 weeks or until complete wound healing, at the dose of 4 µg/cm²/application
  Other Names: BC Very low dose
  Arms: Very Low Dose BioChaperone PDGF-BB

SUMMARY:
This is an open-label, active-control, multicentre, parallel group, randomised and dose-finding efficacy and safety study.

Compare the efficacy and safety of BioChaperone PDGF-BB applied at 12.5 µg/cm² every two days for up to 20 weeks to becaplermin gel (Regranex® Gel 0.01%) applied daily for up to 20 weeks for the treatment of neuropathic diabetic foot ulcer.

Assess the effect of a double dose of BioChaperone PDGF-BB (25 µg/cm²) applied every two days for up to 20 weeks.

DETAILED DESCRIPTION:
After the screening visit, the eligible patient population randomly receive one of the three following topical drugs:

* BioChaperone™ PDGF-BB 12.5 µg/cm²/application for 20 weeks,
* BioChaperone™ PDGF-BB 25 µg/cm²/application for 20 weeks, or
* BioChaperone™ PDGF-BB 4 µg/cm²/application for 20 weeks, or
* Beclapermin gel 6.25 µg/cm²/application for 20 weeks.

The assessment schedule for all the four groups is weekly once (7 day duration) till the 8th week (visit 10) and once in two weeks (14 day duration) thereafter till the end of study. The maximum number of visits expected is 16. The study data is presented at the end of 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 years old or older, with type 1 or 2 diabetes mellitus.
* Single full-thickness plantar ulcer of the extremity (below the malleolus) extending through the epidermis and dermis, but not involving bone, tendons, ligaments or muscles (grade IA as defined by University of Texas Diabetic Wound Classification).
* Chronic ulcer of at least six weeks despite appropriate wound care.
* Ulcer area (greatest length by greatest width), following sharp debridement, of 1 to 10 cm², both inclusive.
* Well controlled infection or cellulitis (systemic antibiotherapy).
* Peripheral neuropathy as assessed by Semmes-Weinstein monofilament test or by the bio esthesimeter (vibration perception threshold).
* Adequate arterial blood supply, to be measured by (color) doppler ultrasonography, ankle brachial pressure index > 0.60, or ankle systolic pressure > 70 mmHg or toe pressure > 30 mmHg. Ankle brachial pressure index should be lower than 1.3 (which is frequently related to medial artery calcification.
* Women surgically sterile, post-menopausal, or agree to practice adequate contraception and have a negative pregnancy test at screening. Non-nursing.
* Signed informed consent before any study procedure.

Exclusion Criteria:

* Ulcer of other cause or origin: electrical, chemical or radiation insult, bedsores, vascular ulcer or Charcot deformities ulcers.
* Active ulcer infection assessed by clinical examination and radiographic if necessary. Presence of necrosis, purulence or sinus tracts that cannot be removed by debridement.
* Active osteomyelitis affecting the area of the target ulcer.
* Poorly controlled diabetes (uncontrolled glycemia: HbA1c ≥ 12%), renal failure (serum creatinine > 3.0 mg/dL), poor nutritional status (albumin < 3.0 g/dL or total protein < 6.5 g/dL).
* Known connective tissue or malignant disease.
* Concomitant treatment with corticosteroids, immunosuppressive agents, radiation therapy, or anticancer chemotherapy.
* Use of investigational drug/device within 30 days.
* Topical application of any advance wound care on this wound (Growth Factor, antiseptics, antibiotics or debriders) within 7 days.
* Vascular reconstruction within 8 weeks. Patients expected to be noncompliant with the protocol (not available for the duration of the trial, treatment or wound care compliance), or felt to be unsuitable by the Investigator for any other reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2010-06; Primary Completion 2011-02 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Incidence of complete wound closure | 20 WEEKS
  Incidence of complete wound closure

SECONDARY OUTCOMES:
Time to achieve complete wound closure | Study duration 20 weeks
  Time to achieve complete wound closure
Percentage reduction in total ulcer surface area at each visit. | Study duration 20 weeks
Incidence of complete wound healing at week 10 | 10 weeks
Safety Safety Measures | Study duration 20 weeks
  1. Treatment emergent adverse events with investigator's assessment of seriousness, severity, duration and relationship to study medication
  2. Wound-related infections
  3. Changes in standard laboratory tests (hematology, biochemistry and detection of antibodies)

CONTACTS AND LOCATIONS:
Overall Officials: T C Raghuram, MD, Phd, Study Director — Medical Director
Locations (7):
- India (7):
  - Vijay Vachharajani Memorial, Rajkot, Gujarat
  - Jain Institute of Vascular sciences, Bangalore, Karnataka
  - Karnataka Institute of Diabetology, Bangalore, Karnataka
  - Lakeshore Hospital & Research Centre Ltd, Kochi, Kerala
  - Joshi Hospital , Maharashra Medical Foundation, Pune, Maharashtra
  - M.V. Hospital for Diabetes, Chennai, Tamil Nadu
  - S.K. Diabetes Research & Education Centre, Kolkata, West Bengal